CLINICAL TRIAL: NCT04336722
Title: A Double-Blind, Randomized, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Odevixibat (A4250) in Children With Biliary Atresia Who Have Undergone a Kasai Hepatoportoenterostomy
Brief Title: Efficacy and Safety of Odevixibat in Children With Biliary Atresia Who Have Undergone a Kasai HPE (BOLD)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Albireo, an Ipsen Company (Industry)
Responsible Party: Sponsor
Organization: Ipsen (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A4250-011; 2019-003807-37 (EudraCT Number); 2024-512086-14-00 (EU CTIS Number)
Record Dates: First submitted 2020-03-27; First posted 2020-04-07 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Biliary Atresia
Keywords: Kasai
MeSH Terms: conditions — Biliary Atresia | interventions — odevixibat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Odevixibat (A4250) (Experimental): Capsules for oral administration once daily for 104 weeks.
  Interventions: Drug: Odevixibat
- Placebo (Placebo Comparator): Capsules for oral administration (to match active) once daily for 104 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Odevixibat — Odevixibat is a small molecule and selective inhibitor of IBAT.
  Arms: Odevixibat (A4250)
Drug: Placebo — Placebo identical in appearance to experimental drug (odevixibat).
  Arms: Placebo

SUMMARY:
Double-blind, randomized, placebo-controlled, Phase 3 study to investigate the efficacy and safety of odevixibat compared to placebo in children with biliary atresia who have undergone a Kasai hepatoportoenterostomy.

DETAILED DESCRIPTION:
Up to 70 sites will be initiated for this study in North America, Europe, Middle East, and Asia Pacific.

ELIGIBILITY:
Inclusion Criteria:

* A male or female patient with a clinical diagnosis of BA
* Age at Kasai HPE ≤90 days
* Eligible to start study treatment within 3 weeks post-Kasai HPE

Key Exclusion Criteria:

* Patients with intractable ascites
* Ileal resection surgery
* ALT ≥10× upper limit of normal (ULN) at screening
* Patients reliant only on total parenteral nutrition, or not able to take study medication orally, at randomization
* Acute ascending cholangitis (patients may be randomized after resolution of acute ascending cholangitis)
* Choledochal cystic disease
* INR >1.6 (the patient may be treated with Vitamin K intravenously; sample may be redrawn and if INR is ≤1.6 at resampling the patient may be randomized)
* Any other conditions or abnormalities, including congenital abnormalities, major cardiac surgery, hepatic, biliary, or GI disease which, in the opinion of the Investigator or Medical Monitor, may compromise the safety of the patient, the integrity of study results, or patient compliance with study requirements
* Weight <3.5kg at randomization

Max Age: 111 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 254 (Actual)
Dates: Start 2020-07-08 (Actual); Primary Completion 2026-06-26 (Estimated); Study Completion 2026-06-26 (Estimated)

PRIMARY OUTCOMES:
Time from randomization to first occurrence of liver transplant, or death | From baseline to Week 104

SECONDARY OUTCOMES:
Proportion of patients with liver transplant | From baseline to Week 104
  Proportion of patients who are alive and have not undergone a liver transplant
Time to onset of any sentinel events | From baseline to Week 104
  Time to onset of any sentinel events
Total bilirubin levels | From baseline to Weeks 13, 26, 52 and 104
  Total bilirubin level after 13, 26, 52, and 104 weeks of study treatment
Serum bile acid levels | From baseline to Weeks 13, 26, 52 and 104
  Serum bile acid level after 13, 26, 52, and 104 weeks of study treatment
Time to pediatric end-stage liver disease (PELD) score >15 | From baseline to Week 104
  Time to pediatric end-stage liver disease (PELD) score >15
Percentage of participants experiencing Adverse Events (AEs) and Serious Adverse Events (SAEs) | From baseline to Week 104
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Percentage of participants with clinically significant changes in Physical Examination | From baseline to Week 104
  Percentage of participants with clinically significant changes in physical examination findings will be reported. The clinical significance will be graded by the investigator.
Percentage of participants with clinically significant changes in Laboratory Parameters (blood chemistry, hematology and coagulation) | From baseline to Week 104
  Percentage of participants with clinically significant change in laboratory parameters (blood chemistry, hematology and coagulation) will be reported. The clinical significance will be decided by the investigator.
Percentage of participants with clinically significant changes in Abdominal Ultrasound findings | From baseline to Week 26 and Week 104
  Percentage of participants with clinically significant change in Abdominal Ultrasound findings will be reported. The clinical significance will be decided by the investigator.

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (66):
- United States (29):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Stanford Children's Health, Palo Alto, California
  - Rady Children's Hospital, San Diego, California
  - UCSF Benioff Children's Hospital San Francisco, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Nemours/Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Miami, Miami, Florida
  - Children's Healthcare of Atlanta - Emory University School of Medicine, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital, Chicago, Illinois
  - Indiana University school of Medicine, Indianapolis, Indiana
  - Johns Hopkins Children's Center, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Michigan Children's Hospital, Ann Arbor, Michigan
  - Children's Mercy Hospital, Kansas City, Missouri
  - Washington University in St. Louis, St Louis, Missouri
  - NYU Grossman school of Medicine, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - NewYork-Presbyterian Morgan Stanley Children's Hospital, New York, New York
  - The Children's Hospital at Montefiore, The Bronx, New York
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - The Children´s Hospital of Philadelphia, Philadelphia, Pennsylvania
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - UT Southwestern Medical Center, Dallas, Texas
  - University of Utah, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (2):
  - Royal Children's Hospital, Parkville
  - The Children´s Hospital at Westmead, Sydney
- UZ Gent, Ghent, Belgium
- Canada (2):
  - CHU Sainte-Justine, Montreal
  - The Hospital for Sick Children, Toronto
- China (2):
  - Guangzhou Women and Children's Medical Center, Guangzhou, Guangdong
  - Children's Hospital of Fudan University, Shanghai
- France (4):
  - Hôpital Femme Mère Enfant, Bron
  - Bicêtre Hospital, Le Kremlin-Bicêtre
  - Jeanne de Flandre Hospital, Lille
  - Necker University Hospital - Enfants malades, Paris
- Germany (4):
  - Charité - Universitätsmedizin Berlin, Berlin
  - University Medical Center Hamburg-Eppendorf UKE, Hamburg
  - Hannover Medical School, Hanover
  - University Children´s Hospital Tuebingen, Tübingen
- Semmelweis Egyetem I.sz Gyermekgyógyászati Klinika, Budapest, Hungary
- Schneider Children´s Medical Center of Israel, Petah Tikva, Israel
- Italy (6):
  - ASST Papa Giovanni XXIII, Bergamo
  - Meyer Children´s University Hospital, Florence
  - University Hospital of Padova, Padua
  - ISMETT - Istituto Mediterraneo per i Trapianti e Terapie ad Alta Specializzazione, Palermo
  - Ospedale Pediatrico Bambino Gesù, Roma
  - Regina Margherita Children´s Hospital, Turin
- Malaysia (2):
  - Hospital Raja Perempuan Zainab II, Kota Bharu
  - University of Malaya Medical Centre, Kuala Lumpur
- University Medical Center Groningen, Groningen, Netherlands
- Starship Child Health, Auckland, New Zealand
- Instytut Pomnik-Centrum Zdrowia Dziecka, Warsaw, Poland
- South Korea (2):
  - Samsung Medical Center, Seoul
  - Seoul National University Children's Hospital, Seoul
- Hospital Universitari Vall d'Hebron, Barcelona, Spain
- National Taiwan University Hospital, Taipei, Taiwan
- Turkey (Türkiye) (3):
  - Hacettepe University Ihsan Dogramaci Childrens Hospital, Ankara
  - Akdeniz University Medical Faculty, Antalya
  - Istanbul University, Istanbul Medical Faculty, Istanbul
- United Kingdom (2):
  - Birmingham Women´s and Children´s Hospital, Birmingham
  - Leeds General Infirmary, Leeds

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of study participants.
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the US and/or EU.
Access Criteria: Further details on Ipsen's sharing criteria and process for sharing are available here (https://www.ipsen.com/science/clinical-trials/clinical-data-transparency/).
URL: https://www.ipsen.com/science/clinical-trials/clinical-data-transparency/